CLINICAL TRIAL: NCT05442827
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Phase II/III Clinical Study to Explore the Optimal Therapeutic Dose of SHR7280 Tablets and the Efficacy and Safety of SHR7280 Tablets in Subjects With Menorrhagia for Uterine Fibroids
Brief Title: A Phase II/III Study of Efficacy and Safety of SHR7280 Tablets in Subjects With Menorrhagia With Uterine Fibroids
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR7280-301
Record Dates: First submitted 2022-06-16; First posted 2022-07-05 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Uterine Fibroids With Menorrhagia

STUDY DESIGN:
Intervention Model Description: Phase one：300mg/400mgSHR7280 tablets were compared with placebo Phase two：SHR7280 monotherapy group, SHR7280 reverse therapy group and placebo group were controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: SHR7280 tablets (Experimental)
  Interventions: Drug: SHR7280 tablets
- Treatment group B:SHR7280 tablets (Experimental)
  Interventions: Drug: SHR7280 tablets
- Treatment group C:Intervention: Drug: PlaceboSHR7280 tablets blank preparation (Placebo Comparator)
  Interventions: Drug: PlaceboSHR7280 tablets blank preparation

INTERVENTIONS:
Drug: SHR7280 tablets — SHR7280 tablets 300mg for 12 weeks
  Arms: Treatment group A: SHR7280 tablets
Drug: SHR7280 tablets — SHR7280 tablets 400mg for 12 weeks
  Arms: Treatment group B:SHR7280 tablets
Drug: PlaceboSHR7280 tablets blank preparation — Placebo group: SHR7280 tablets blank preparation for 12 weeks
  Arms: Treatment group C:Intervention: Drug: PlaceboSHR7280 tablets blank preparation

SUMMARY:
Phase II:To explore the optimal effective dose of SHR7280 tablets in subjects with menorrhagia with uterine fibroids as a phase III treatment dose.

Phase III:To evaluate the efficacy of the selected dose of SHR7280 compared with placebo in reducing menstrual bleeding in subjects with menorrhagic uterine fibroids in phase II studies.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent has been signed and dated;
2. Non-menopausal women between the ages of 18 and 49 (including 18 and 49);
3. Single or multiple uterine fibroids were confirmed by ultrasound examination during screening, and the maximum diameter of at least one fibroid was ≥2 cm;
4. Heavy menstrual bleeding measured by the alkaline hematin method during screening;
5. 3 months before screening, the subject's menstrual cycle is 21-38 days, and the period is no more than 14 days;
6. The pregnancy test was negative on the day of screening visit and randomization;
7. Human papillomavirus (HPV) testing should be added for subjects who have cervical cytology at the time of screening visit and whose TCT results are atypical squamous cells (ASC-US) of uncertain significance, or who test negative for high-risk HPV.

Exclusion Criteria:

1. Excessive menstrual bleeding and anemia caused by other reasons;
2. A history of depression or clinically significant depression;
3. Have a history of drug abuse, drug dependence;
4. History of smoking and alcohol abuse within 3 months prior to screening;
5. A history of delivery, breastfeeding and miscarriage within 6 months prior to screening;
6. Patients who received myomectomy within 3 months before screening, and patients who received uterine artery embolization, or high intensity focused ultrasound (HIFU) ablation within 6 months before screening;
7. Patients who underwent endometrial resection within 1 year prior to screening;
8. Patients with severe infection (one organ or whole body infection caused by pathogenic microorganism, and failure or death of the organ or multiple organs caused by infection), severe trauma (ISS ≥16 points) or major surgery (grade III/IV surgery in Surgical Classification Catalogue) within 6 months prior to screening;
9. Previous clinical major systemic disease, endocrine or metabolic abnormalities;
10. Having past or current thromboembolic disease or having a risk factor for thromboembolic disease (stage 2 only);
11. Previous history of malignant tumors such as ovary, breast, uterus, liver, hypothalamus and pituitary gland;Known or suspected sex hormone-dependent malignancies;
12. Any pre-existing disease or symptom (e.g., chronic intestinal disease, Crohn's disease, ulcerative colitis) that may affect systemic functioning of the body and may affect absorption, excessive accumulation, metabolism, or change the excretion pattern of the test drug;
13. Persons with prior known serious mental illness or inability to understand the purpose, methods, etc. of the clinical trial, and who did not follow the study procedures;
14. Live (attenuated) vaccine (other than influenza vaccine) received within 1 month prior to screening or planned during the trial;
15. Other reasons that the investigator considered inappropriate for participation in the study.
16. Follicle-stimulating hormone (FSH) ≥25U/L during screening;
17. Hb < 6 g/dL during screening;
18. Moderate to severe liver impairment during screening, including aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin (unless Gilbert's diagnosis is known) ≥2.0 times the upper limit of the reference range;
19. During screening, endometrial biopsy should be performed if endometrial thickness > 18 mm is indicated by gynecological ultrasound or if the investigator deems it necessary. Endometrial histological abnormalities indicated by endometrial biopsy should be performed (only in the first stage).
20. Active pelvic inflammatory disease (PID) during screening;
21. QTcF≥450ms during screening;
22. Infectious disease screening resultshave clinical significance;
23. 6 months before enrollment, endometrial biopsy revealed significant endometrial histological abnormalities;If the subject has no sexual life history or the investigator determines that it is not necessary, the subject may be exempted (stage 2 only);
24. Two or more blood transfusions within 9 months prior to enrollment, or requiring transfusion therapy within 2 months prior to enrollment, or having any condition requiring immediate transfusion;
25. 1 month before admission, she used any drugs that inhibited or induced liver metabolism of drugs (liver drug enzyme inhibitors such as chloramphenicol, allopurinol,ketoconazole, fluoroquinolones, etc., and liver drug enzyme inducers such as carbamazepine, dexamethasone, phenobarbital, phenytoin sodium, rifamequine);
26. Participants in and enrolled in clinical trials of any drug or medical device within 3 months prior to enrollment, or who were still in the follow-up period of a clinical study or within 5 half-lives of the tested drug prior to screening, whichever is longer.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 357 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Phase one：Percentage of subjects with menstrual bleeding < 80 mL and a reduction of ≥50% from baseline | After treatment at week 12
Phase two：Percentage of subjects with menstrual bleeding < 80 mL and a reduction of ≥50% from baseline | After treatment at week 24

SECONDARY OUTCOMES:
Percentage of subjects with menstrual bleeding < 80 mL and a reduction of ≥50% from baseline（Phase one） | The treatment ended at week 4 and 8
percentage of subjects without menstrual bleeding or spotting （Phase one） | The treatment ended at week 4, 8 and 12
Changes in hemoglobin concentration from baseline（Phase one） | The treatment ended at week 4, 8 and 12
Changes in uterine volume and maximum fibroid volume from baseline（Phase one） | The treatment ended at week 8 and 12
patient global impression of change scale evaluation，The minimum is 1, the maximum is 7, and higher scores mean worse results（Phase one） | The treatment ended at week 12
Changes in uterine fibroid symptoms from baseline（Phase one） | The treatment ended at week 12
Changes in health related Quality of Life Questionnaire (UFS-QOL) scores from baseline，The minimum is 37 and the maximum is 185, with higher scores indicating worse results（Phase one） | The treatment ended at week 12
Number of Participants with Adverse events（Phase one） | Stage ⅱ ended, about 30 weeks
The interval between stopping the medication and resuming menstruation（Phase one） | Stage ⅱ ended, about 30 weeks
The amount of menstrual bleeding when the medication was stopped until menstruation resumed（Phase one） | Stage ⅱ ended, about 30 weeks
Number of days of menstruation from the time of discontinuation of the medication to the time of resumption of menstruation(Phase one) | Stage ⅱ ended, about 30 weeks
SHR7280 concentration in plasma(Phase one) | Before and at week 4, 8 and 12 after administration
Serum concentrations of estradiol, luteinizing hormone, follicle stimulating hormone and progesterone(Phase one) | Before and at week 4, 8 and 12 after administration
Percentage of subjects with menstrual bleeding < 80 mL and a reduction of ≥50% from baseline（Phase two） | At the end of weeks 4,8,12,16,20,28,32,36,40,44,48,52
Changes in menstrual bleeding from baseline were assessed using the Alkaline hematin method (AH)（Phase two） | At the end of weeks 4,8,12,16,20,24,28,32,36,40,44,48,52
percentage of subjects without menstrual bleeding or spotting (Phase two) | Weeks 4,8,12,16,20,24,28,32,36,40,44,48,52
change in Hb concentration from baseline (Phase two） | The treatment ended at 4, 8, 12, 16, 20, 24, 36, 44, 52 weeks
Changes in uterine volume and maximum fibroid volume from baseline(Phase two) | The treatment ended at weeks 12, 24, and 52
patient global impression of change scale evaluation，The minimum is 1, the maximum is 7, and higher scores mean worse results(Phase two) | The treatment ended at weeks 12, 24, and 52
Changes in health related Quality of Life Questionnaire (UFS-QOL) scores from baseline，The minimum is 37 and the maximum is 185, with higher scores indicating worse results(Phase two) | The treatment ended at weeks 12, 24, and 52
Number of Participants with Adverse events(Phase two) | Stage ⅲ ended at about 74 weeks
The interval between stopping the medication and resuming menstruation(Phase two) | Stage ⅲ ended at about 74 weeks
The amount of menstrual bleeding when the medication was stopped until menstruation resumed(Phase two) | Stage ⅲ ended at about 74 weeks
Number of days of menstruation from the time of discontinuation of the medication to the time of resumption of menstruation(Phase two) | Stage ⅲ ended at about 74 weeks
plasma SHR7280 concentration data(Phase two) | Treatment ended at 4, 24, 36, 52 weeks before administration
serum E2, LH, FSH and P concentrations at each point of view(Phase two) | Treatment was completed at 4, 8, 12, 16, 20, 24, 36, 44, 52 weeks before administration

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided